CLINICAL TRIAL: NCT05412771
Title: Bases Évolutives Et Fonctionnelles De La Menstruation Chez Les Femmes - 2
Brief Title: Evolutive and Functional Bases of Menstruation in Women - 2
Acronym: EVOMENS-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: C21-20; 2021-A02779-32 (Registry Identifier: IDRCB)
Record Dates: First submitted 2022-05-23; First posted 2022-06-09 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Menstruation
Keywords: endometrium; comparative genomics
MeSH Terms: interventions — Hysteroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Main cohort (Experimental): This is a single-arm study. Samples are collected from consenting donors undergoing surgery for medical purposes.
  Interventions: Procedure: Hysteroscopy

INTERVENTIONS:
Procedure: Hysteroscopy — Samples will be collected from consenting patients undergoing a surgical hysteroscopy for medical purposes

SUMMARY:
Menstruation corresponds to the shedding of the uterine lining when fecundation has not occurred. This is a recent evolutionary innovation in primates, and the cellular and genetic changes that led to the acquisition of menstruation are not well understood. Additionally, the uterine lining is poorly characterized in humans across the menstrual cycle, which hinders both evolutionary and medically-relevant analyses.

In this study, the research team are collecting uterine endometrial tissue samples from female donors undergoing uterine surgery for benign conditions, to profile gene expression and gene regulatory elements in the major cell types that compose the uterine lining during the secretive phase of the menstrual cycle. The investigators will compare this data to similar samples collected from other primates at the same time point in the female hormonal cycle.

The objective is to identify genes that have acquired novel regulation and/or expression patterns and which may be involved in menstruation, as well as better characterize the cellular and molecular pathways at work in the uterine lining of women for translational medicine purposes.

DETAILED DESCRIPTION:
Collection:

The research team will collect endometrial biopsies or discarded tissue scraps from medical practice from 20 consenting female donors undergoing surgical hysteroscopy for benign uterine conditions.

Primary objective:

The research team will perform transcriptome sequencing and open chromatin profiling from the tissue samples and compare to similar data produced from non-human primates that either do or do not menstruate. They will identify and characterize genes and non-coding regulatory elements differentially used in menstruating species and involved in the evolution of menstruation.

Secondary objectives:

The research team will profile and characterize non-coding RNAs expressed in the human endometrium.

The research team will establish 3D cell cultures (organoids) from the tissue samples for further functional validations of the primary objective.

ELIGIBILITY:
Inclusion Criteria:

* Be between 18 and 50 years old.
* Have mensturation at the time of their participation
* Have given their written consent
* Have an indication for surgery of hysteroscopy for removal of a polyp and/or fibroid and/or endometrial, endometrialctomy for presumed benign pathology and/or management of a uterine malformation, scheduled between days 21 and 25 of their menstrual cycle
* Covered by social security

Exclusion Criteria:

* Using an intrauterine device contraceptive method during the study or within the previous three months
* To be Pregnant at the time of collection
* Have been pregnant in the three months prior to collection
* Have had amenorrhoea in the three months prior to collection
* Have received hormonal treatment within the three months prior to collection
* Have participated in a clinical study within 3 months prior to collection
* Have a personal history of breast, ovarian, body or cervical cancer
* Have a diagnosis of endometriosis
* Have a diagnosis of adenomyosis
* Have a diagnosis of Lynch syndrome
* Undergoing hysteroscopy for a condition other than those listed in the inclusion criteria
* Women who have not given written consent
* Women who are breastfeeding
* Women with a body mass index (BMI) of less than 18.5 or more than 30

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2022-11-23 (Actual); Primary Completion 2026-05-23 (Estimated); Study Completion 2027-10-25 (Estimated)

PRIMARY OUTCOMES:
Transcriptomics | 18 months
  Characterisation of genes involved in the evolutionary establishment of menstruation: transcriptome sequencing and identification of genes differentially expressed between menstruating and non-menstruating species in each cell type using DeSEQ analysis (FDR-corrected p-value < 0.05)
Open chromatin analysis | 18 months
  Characterisation of non-coding regulatory elements specifically involved in the evolutionary establishment of menstruation: open chromatin sequencing (ATAC-seq) and identification of non-coding genomic regions differentially activated between menstruating and non-menstruating species in each cell type using DeSEQ analysis (FDR-corrected p-value < 0.05)

SECONDARY OUTCOMES:
Non-coding transcriptomics | 18 months
  Characterisation of non-coding transcripts expressed in the endometrium in menstruating and non-menstruating species in each cell type by transcriptome sequencing, transcript assembly and annotation of expressed non-coding transcripts in each genome
3D cell culture - establishment | 18 months
  Obtaining 3D cell cultures ("organoids") to validate the observations of the main objective: proliferation and expansion time-course assessed by bright-field microscopy
3D cell culture - structural evaluation | 18 months
  Topographical evaluation of the 3D cell cultures with H/E and PAS staining
3D cell culture - cell types evaluation | 18 months
  Profiling of characteristic cell markers in the 3D cell cultures via immunochemistry and immunofluorescence staining (MUC1, Cytokeratin7, EPCAM, Vimentin, CD13, ESR, PGR)
3D cell culture - gene expression | 18 months
  Gene expression profiling of the 3D cell cultures by PCR to compare to the transcriptomes from fresh tissues.

CONTACTS AND LOCATIONS:
Locations (1):
- Pitié salpétrière, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Data generated from tissue samples from donors who gave expressed consent will be shared in the European Genome-Phenome Database (EGA).
Supporting Information: Study Protocol, CSR, Analytic Code